CLINICAL TRIAL: NCT00463736
Title: Magnesium Sulfate Versus Placebo for Tocolysis in Preterm Premature Rupture of Membranes
Brief Title: Magnesium Sulfate Versus Placebo for Tocolysis in PPROM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment proceeding too slowly
Sponsor: Regional Obstetrical Consultants (Other)
Responsible Party: Principal Investigator, Lorrie Mason, Christian Briery MD, Regional Obstetrical Consultants
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-006
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Preterm Premature Rupture of Membranes
Keywords: short term tocolysis; preterm premature rupture of membranes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Magnesium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium sulfate (Active Comparator): x 48 hours IV
  Interventions: Drug: Magnesium sulfate
- Normal saline (Placebo Comparator): x 48 hours IV
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate

SUMMARY:
Study compares the outcomes of women between 26 and 32 wks gestation with rupture of membranes. Women randomized to receive tocolysis with magnesium sulfate x 48 hrs or placebo of saline IV x 48 hrs. Antibiotics and antenatal steroids given to both groups.

DETAILED DESCRIPTION:
The majority of studies of the effectiveness of tocolysis with PPROM were in the 1980s prior to the commmon usage of antenatal steroids and prophylactic maternal antibiotics. In most studies, tocolysis was not attempted prior to the onset of labor in this group of women. The ACOG Practice Bulletin of June 1998 concedes that the recommendation of tocolysis to permit administration of steroids and maternal antibiotics is based primarily upon consensus, not consistent scientific evidence.

The purpose of this study, which will randomize 128 subjects to tocolysis or no tocolysis, is to prospectively assess whether short term (48 hr) tocolysis affords benefit to women and babies between 26 and 32 weeks gestation with PPROM.

Subjects will be enrolled at 1-2 high risk hospitals in Chattanooga and Knoxville. All English and Spanish speaking women 18-45 years with PPROM and cervical dilation <4 will be eligible. Women with suspected intrauterine infection, positive fetal lung maturity, or > 6 hours tocolysis at time of admission will be excluded.

Both groups of women will receive continuous fetal monitoring, antibiotics, and antenatal steroids (if not previously administered). Both groups will be evaluated every 2-4 hours for fetal and maternal well being. Both groups will receive IVF at 125cc/hr, and the treatment group will be loaded with 4 grams of magnesium sulfate and receive maintainence dose of 2 grams/hr x 48 hrs.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* preterm premature rupture of membranes
* 26 - 32.6 weeks gestation
* cervical dilation </= 4 cm

Exclusion Criteria:

* suspected intrauterine or intraamniotic infection
* > 6 hours of tocolysis prior to admission
* positive fetal lung maturity

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2007-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
hours of latency to delivery | 0 hours to > 168 hours
  from start of study drug to delivery

SECONDARY OUTCOMES:
maternal postpartum length of stay | 0 hours to > 168 hours
  from start of study drug to delivery
maternal infection rates | 0 hours to > 168 hours
  from start of study drug to maternal discharge from hospital
neonatal ventilator days | 0 to 28 days
  from delivery to 28 days of life
neonatal early onset infection | 0 to 28 days
  from delivery to 28 days of life
neonatal length of stay | 0 to 28 days
  from delivery to 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Christian M Briery, MD, Principal Investigator — Regional Obstetrical Consultants; UT Chattanooga OB-GYN Department
Locations (1):
- Regional Obstetrical Consultants, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046